CLINICAL TRIAL: NCT05240170
Title: Retrograde Intrarenal Surgery for Treatment of Stones in Congenital Anomalous Kidneys: Case Matched Comparative Study With Extracorporeal Shockwave Lithotripsy
Brief Title: RIRS for Treatment of Stones in Congenital Anomalous Kidneys
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Al-Azhar University (Other)
Responsible Party: Principal Investigator, Abul-fotouh Ahmed, Professor, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Uro_Azhar_1_022
Record Dates: First submitted 2022-02-04; First posted 2022-02-15 (Actual); Last update posted 2022-04-26 (Actual); Status verified 2022-04

CONDITIONS: Renal Calculi; Renal Anomaly
MeSH Terms: conditions — Kidney Calculi

STUDY DESIGN:
Intervention Model Description: The 1st group: RIRS The 2nd group: SWL
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- RIRS group (Experimental): The standard RIRS will be performed using a disposable flexible ureteroscope. Holmium: YAG laser will be used for stone dusting and fragmentation. If indicated, JJ ureteral stent will be placed at the end of the procedure.
  Interventions: Device: RIRS
- SWL group (Experimental): The medical records of all patients who underwent SWL at our institution in the past five years will be reviewed. Patients with renal rotation or position anomalies, as defined by NCCT and/or IVU, will be included for possible study participation.
  Interventions: Device: SWL

INTERVENTIONS:
Device: RIRS — The standard RIRS will be performed using a disposable flexible ureteroscope. Holmium: YAG laser will be used for stone dusting and fragmentation. If indicated, JJ ureteral stent will be placed at the end of the procedure.
  Other Names: Retrograde flexible ureteroscopy
  Arms: RIRS group
Device: SWL — Patients who underwent SWL at our institution in the past five years. According to (a) the type of renal anomaly (rotation, position, or rotation/position anomaly), (b) the size of the stone (±5 mm), (c) location of the stone (lower polar or non-lower polar), and (d) density of the stone (>800 HU or ≤800 HU), matched cases will be selected for comparison.
  Arms: SWL group

SUMMARY:
The anatomic renal abnormalities like altered spatial relations with adjacent organs, abnormal calyceal orientation, and anomalous vascular patterns make the active treatment of stones in the congenitally malformed kidney a great challenge for urologists. In this prospective study, the investigators will evaluate the outcome of retrograde intrarenal surgery (RIRS) with extracorporeal shockwave lithotripsy (SWL) for the treatment of stones in the kidneys with rotation or position anomalies.

DETAILED DESCRIPTION:
In current stone guidelines, the recommendations for stone therapy in the kidneys with normal anatomy are clearly stated; however, there is also no clear suggestion and treatment modality in regards to the stone treatment in anomalous kidneys. Nowadays, open surgery, percutaneous nephrolithotomy (PNL), SWL, and RIRS are used for the treatment of these kidney stones. However, there is no clear consensus on which treatment modalities should be used; each modality has its unique advantages and drawbacks. in this study, the investigators will prospectively evaluate the safety and efficacy of RIRS in treatment of stones in kidneys with rotation or position anomalies. The investigators will compare the results with a matched group of patients who were treated with SWL. The results of this study may help clarify treatment options in the management of patients with stones and renal anomalies.

ELIGIBILITY:
Inclusion Criteria:

* The study will include patients with renal stones up to 20 mm in size in a kidney with rotation or position anomalies.

Exclusion Criteria:

* Pregnant women.
* Uncorrectable coagulation disorders.
* Urinary tract obstruction distal to the stone.
* Active infection.
* Stone in a calyceal diverticulum

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 160 (Estimated)
Dates: Start 2022-03-15 (Actual); Primary Completion 2024-02-15 (Estimated); Study Completion 2024-07-15 (Estimated)

PRIMARY OUTCOMES:
Stone-free rate | 3-months after the intervention.
  Stone-free status is defined as no residual fragments of ≥3 mm on abdominal NCCT and/or X-ray KUB.

SECONDARY OUTCOMES:
Complication rate | intraoperative till 3 months postoperative complications
  intraoperative and postoperative complications
operative time | the procedure time
  from starting till the end of the procedure
Re-treatment rate | during the post-operative 3 months
  need for reintervention

CONTACTS AND LOCATIONS:
Overall Officials: Abul-fotouh Ahmed, MD, Principal Investigator — Al-Azhar University Hospitals, Cairo, Egypt
Locations (1):
- Urology Department, Al-Azhar University Hospital, Cairo, Egypt